CLINICAL TRIAL: NCT03806049
Title: ENGOT-OV42 / NSGO-AVATAR: A Three-arm Randomized Study to Evaluate the Efficacy of Niraparib-bevacizumab-dostarlimab Triplet Combination Against Niraparib-bevacizumab Doublet Combination and Against Standard of Care Therapy in Women With Relapsed Ovarian Cancer Where Platinum Combination Therapy is an Option.
Brief Title: Trial Comparing Niraparib-bevacizumab-Dostarlimab and Niraparib-bevacizumab to Standard of Care in Recurrent Ovarian Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of financial support
Sponsor: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENGOT-OV42 / NSGO-AVATAR
Record Dates: First submitted 2019-01-13; First posted 2019-01-16 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2019-09

CONDITIONS: Ovarian Cancer
Keywords: chemotherapy-free regimen; niraparib; bevacizumab; dostarlimab; recurrent ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib; Bevacizumab; dostarlimab; Carboplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: randomized, open-label, three arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A: triplet (Experimental): chemotherapy-free combination of niraprib + bevacizumab + Dostarlimab
  Interventions: Drug: Niraparib; Drug: Bevacizumab; Drug: TSR042
- B: Doublet (Experimental): chemotherapy-free combination of niraparib + bevacizumab
  Interventions: Drug: Niraparib; Drug: Bevacizumab
- C: standard of care (Active Comparator): Standard of care chemotherapy: Carboplatin + paclitaxel
  Interventions: Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Niraparib — given orally once daily
  Other Names: Zejula
  Arms: A: triplet; B: Doublet
Drug: Bevacizumab — given as iv infusion every three weeks
  Other Names: Avastin
  Arms: A: triplet; B: Doublet
Drug: TSR042 — Given as IV infusion every three weeks
  Arms: A: triplet
Drug: Carboplatin — given as iv infusion every three weeks
  Arms: C: standard of care
Drug: Paclitaxel — given as iv infusion every three weeks
  Arms: C: standard of care

SUMMARY:
ENGOT-OV42 / NSGO-AVATAR: This three-arm randomized trial is to demonstrate efficacy of niraparib-bevacizumab-dostarlimab triplet combination against standard of care treatment and to demonstrate efficacy of niraparib-bevacizumab-dostarlimab triplet combination against niraparib-bevacizumab doublet combination for patients with platinum-sensitive epithelial ovarian, fallopian tube, or peritoneal cancer

DETAILED DESCRIPTION:
This is a multicenter randomized open-label trial to compare two different chemotherapy-free arms against standard of care treatment in patients with recurrent ovarian cancer with >6 months of chemotherapy-free interval to prior therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent platinum-sensitive epithelial ovarian, fallopian tube, or peritoneal cancer (platinum sensitivity defined as no recurrence within 6 months of last receipt of platinum/chemotherapy).
2. High-grade serious or high-grade endometrioid histology or any histology with known BRCA mutation.
3. Patient consents to perform BRCA test, and PD-L1 expression.
4. Prior line of therapy: Patients must have received platinum-containing therapy for primary disease.
5. No limits on number of platinum-based therapies.
6. Up to one non-platinum-based line of therapy in recurrent setting is allowed.
7. Patients may have received bevacizumab (or other anti-VEGF therapy) prior to entering in the trial.
8. Patients may have participated in a PARP inhibitor maintenance trial or have received maintenance PARP inhibitor therapy are allowed, though it is necessary to unblind patient in order to correctly stratify. Patients who received a PARP inhibitor as definitive are not eligible. Patients may have participated in a trial containing immune-checkpoint inhibitor.
9. Target group: Age 18+
10. Histological confirmed ovarian, fallopian tube or peritoneal cancers
11. Patients must give informed consent
12. Patients may have undergone primary or interval debulking surgery
13. Patients may have received bevacizumab or other anti-angiogenic therapy
14. Patients may have received a PARP inhibitor as first-line maintenance therapy.
15. Patients must have disease that is measurable according to RECIST or assessable according to the GCIG criteria
16. The patient agrees to complete PROs (QoL questionnaire) during study treatment AND at one additional time point 8 weeks following progression of disease
17. ECOG performance status 0-2
18. Adequate organ function

    1. Absolute neutrophil count (ANC) ≥1,5 x 109/L
    2. Platelets >100 x 109/L
    3. Hemoglobin ≥ 9g/dl
    4. Serum creatinine ≤1.5x upper limit of normal (ULN) or calculated creatinine clearance ≥50mL/min using Cockcroft-Gault formula
    5. Total bilirubin ≤1.5x ULN
    6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5x ULN unless liver metastases are present, in which case they must be ≤5x ULN.
19. Able to take oral medications
20. Life expectancy of at least 12 weeks
21. Patients must fulfill all inclusions criteria and according to investigator fit to receive niraparib, bevacizumab and TSR042.
22. Women of childbearing potential must use adequate birth control for the duration of study participation -

Exclusion Criteria:

Ovarian sarcomas, small cell carcinoma with neuroendocrine differentiation, non-epithelial cancers and cancer types not mentioned in the inclusion criteria 2. Concurrent cancer therapy 3. Concurrent treatment with an investigational agent or participation in another clinical trial 4. Major injuries or surgery within the past 21 days prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period 5. Previous malignant disease: patients are not eligible for the study if diagnosis, detection or treatment of invasive cancer (other than ovarian cancer; with the exception of basal or squamous cell carcinoma of the skin that was definitively treated) was detected within 2 years prior to randomization 6. Active infections or other serious underlying significant medical illness, abnormal laboratory finding or psychiatric illness/social situation that would, in the Investigator's judgment, makes the patient inappropriate for this study 7. Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug 8. History of bowel obstruction, including sub-occlusive disease, related to the underlying disease and history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess. Evidence of recto-sigmoid involvement by pelvic examination or bowel involvement on CT scan or clinical symptoms of bowel obstruction 9. Known contraindications to PARP inhibitors, VEGF directed therapy or immune checkpoint inhibitors 10. Known uncontrolled hypersensitivity to the investigational drugs 11. History of major thromboembolic event defined as:

* Uncontrolled pulmonary embolism (PE)
* Deep venous thrombosis (DVT)
* Other related conditions, though patients with stable therapeutic anticoagulation for more than three months prior randomization are eligible for this study. This also apply to PE & DVT.

  12. History of a cerebral vascular accident, transient ischemic attack or subarachnoid hemorrhage within the past 3 months 13. History of clinically significant hemorrhage in the past 3 months 14. Uncontrolled and/or symptomatic CNS metastasis or leptomeningeal carcinomatosis (Dexamethasone/prednisone therapy will be allowed if administered as stable dose for at least one month prior randomization) 15. Significant cardiovascular diseases, including uncontrolled hypertension, clinically relevant cardiac arrhythmia, unstable angina or myocardial infarction within 6 months prior to randomization, congestive heart failure > NYHA III, severe peripheral vascular disease, QT prolongation >470 msec ,clinically significant pericardial effusion 16. Pregnancy or breastfeeding. Patients with preserved reproductive capacity, unwilling to use a medically acceptable method of contraception for the duration of the trial and for 3 months afterwards.

  17. Radiographic evidence of cavitation or necrotic tumors with invasion of adjacent major blood vessels 18. Active or chronic hepatitis C and/or B infection 19. Persistence of clinically relevant therapy related toxicity from previous chemotherapy 20. Proteinuria as demonstrated by: (a) urine protein: creatinine (UPC) ratio >/= 1.0 at screening OR (b) urine dipstick for proteinuria >/=2+ (patients discovered to have >/=2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hr urine collection and must demonstrate </=1g of protein in24 hours to be eligible 21. Patients must not have any known history of MDS 22. Patients must not have known persistent (> 4 weeks) ≥ Grade 2 hematological toxicity from prior cancer therapy 23. Patients must not have known ≥ Grade 3 thrombocytopenia or anemia with the last chemotherapy regimen.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 42 months
  the time from randomization until the date of the first objective radiological disease progression according to investigator assessment of RECIST v1.1 or death by any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression Free Survival in Sub-Population in months | 42 months
  the time from randomization until the date of the first objective radiological disease progression according to investigator assessment of RECIST v1.1 or death by any cause, whichever occurs first for the predefined study subgroups.
Progression Free Survival 2 in each group according to trial stratification factors | 58 months
  The time from randomization until date of second objective radiological disease progression according to investigator assessment of RECIST v1.1 or death by any cause, whichever occurs first for the predefined study subgroups
TFST (Time to First Subsequent Therapy) | 44 months
  The time from randomization until date of subsequent cancer therapy
TSST (Time to Second Subsequent Therapy) | 60 months
  The time from randomization until date of second subsequent cancer therapy
Overall survival (OS) | 72 months
  The time from randomization until date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: MANSOOR RAZA R MIRZA, Study Chair — NSGO
Locations (8):
- Denmark (4):
  - NSGO, Copenhagen, Region Sjælland
  - Rigshospitalet, Copenhagen, Region Sjælland
  - Rigshospitalet, København Ø, Region Sjælland
  - Aalborg University Hospital, Aalborg
- Tampere University Hospital, Tampere, Finland
- Norway (3):
  - Haukeland University Hospital, Bergen, Haukeland
  - Norwegian Radium Hospital, Oslo
  - The Norwegian Radium Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No
All individual participant data will be anonymized